CLINICAL TRIAL: NCT06288126
Title: Evaluation of Clinical and Ecographic Risk Markers in Pregnancies at High and Low Risk for the Development of Glycemic and Metabolic Complications in Pregnancy
Brief Title: Maternal and Fetal Metabolic Changes
Acronym: MoMM-FET
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Tommaso Simoncini, Full Professor, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: MoMM-FET
Record Dates: First submitted 2024-02-06; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy Related; Maternal-Fetal Relations; Metabolism Disorder, Glucose
Keywords: metabolism; insulin resistance; adipose tissue; insulin-signalling pathway
MeSH Terms: conditions — Glucose Metabolism Disorders; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk Group: This group include women at high risk for gestational diabetes (GDM) according to most of the European guidelines. They have one or more of the following criteria: age ≥35 years, overweight or obesity, family history of diabetes, high-risk ethnicities, history of previous GDM or previous macrosomia, and high levels of fasting glycemia during the first trimester screening.
- Low Risk Group: This group will include women at low risk for GDM according to most of the European guidelines. They have none of the following criteria: age ≥35 years, overweight or obesity, family history of diabetes, high-risk ethnicities, history of previous GDM or previous macrosomia, and high levels of fasting glycemia during the first trimester screening.

SUMMARY:
The goal of this observational prospective project is to study the metabolic alterations during normal and complicated pregnancies, obtaining an early detection of metabolic changes, offering new insights into future prevention and treatment strategies for both mother and offspring.

Primary objectives:

* measurement of maternal blood adipokine levels, during the first trimester of pregnancy, in two groups of women (high and low risk), in order to identify early markers which, in conjunction with the medical history, can identify women at increased risk of developing GDM
* ultrasound measurement of adipose tissue deposits at ectopic sites, comparing low- and high-risk women, and assessing the effect of pregnancy on these deposits.
* Identification, by targeted ultrasound assessment, of fetuses at increased risk of macrosomia.

Secondary objectives:

* Evaluation of the prevalence of GDM and its complications in a population of low- and high-risk women.
* Evaluation of neonatal complications in children born to low- and high-risk mothers (need for resuscitation, hypoglycaemia, hypocalcaemia, admission to neonatal intensive care unit).

The participants will be recruited during first trimester ultrasound after signing the informed consent.

DETAILED DESCRIPTION:
Pregnancy has been defined "a stress test for life". During pregnancy, even if uncomplicated, women experience metabolic and cardiovascular changes that predispose to vascular endothelial dysfunction. Women who are already predisposed to this phenotype develop gestational hypertension or gestational diabetes (GDM), which can re-emerge later in life. This has been demonstrated by several studies in which the presence of pregnancy diseases (GDM, maternal preeclampsia and fetal growth disorder) correlate with the development of chronic disorders, such as chronic hypertension, diabetes mellitus and metabolic syndrome, suggesting a common pathogenic pathway. From this point of view, pregnancy constitutes a unique period to evaluate metabolic and cardiovascular markers, to better understand the pathogenesis of these disorders and possibly obtain preventive strategies. The identification of early biomarkers of metabolic dysfunction would be particularly useful in overweight and obese pregnant women. There is a growing prevalence of obesity worldwide; in developed Countries, 40-50% of the pregnant population is overweight and obese, which is, according to a recent report from the United Kingdom, the main contributing cause of death during gestation.

In addition, obesity and maternal hyperglycaemia during pregnancy may induce intrauterine overnutrition and fetal hyperinsulinemia, resulting in excessive fetal growth. Fetal macrosomia is associated with an increased risk of perinatal morbidity and mortality. Large babies have increased risk of intrapartum complications such as prolonged labour and shoulder dystocia. Moreover, the environmental and metabolic characteristics of intrauterine life deeply influence the individual in the long-term as a child and through adulthood, with possible adverse metabolic consequences, including predisposition to insulin resistance and obesity.

The evaluation of fetal tissue distribution and the recently introduced study of the fetal liver volume constitute very interesting markers of fetal adiposity and could be used as early indicators of insulin resistance in newborns.

The participants will be recruited during first trimester ultrasound after signing the informed consent. At 11-13 weeks:

* Ultrasound evaluation of fetal biometry and amniotic fluid will be performed. Periodic maternal anthropometric evaluation (weight gain and body mass index (BMI), blood pressure). Women will be divided in lean, overweight and obese.
* Blood sample for inflammatory cytokines will be taken.
* Maternal body composition evaluation through bioimpedance and/or highly reliable ultrasound-based analysis of ectopic fat. This approach is ideal to provide biomarkers of insulin resistance. In brief, women will be evaluated by a standardized set of US clips for the assessment of liver fat, cardiac fat, abdominal subcutaneous and visceral fat.

At 16-18 weeks: standard screening for gestational diabetes for high risk women, as for clinical practice

At 24-28 weeks:

* Standard screening for gestational diabetes to all women
* Fetal ultrasound to study fetal liver volume and/or subcutaneous fat tissue quantification. These constitute innovative techniques to obtain an early identification of macrosomic fetuses.

At delivery:

* Information on mode of delivery and any complications
* Within 48 hours of birth, anthropometric assessment of the infant according to clinical practice (weight, abdominal and head circumference).

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* first visit between 11 and 14 weeks of pregnancy

Exclusion Criteria:

* consent withdrawal
* multiple pregnancy
* prepregnancy diabetes mellitus
* women undergoing therapy with oral hypoglycaemic drugs
* previous bariatric surgery
* fetal chromosomal and/or major structural abnormalities were excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a singleton pregnancy attending our Centre for aneuploidies screening in the first trimester.
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Blood adipokine levels | Between 11 (+0 days) and 13 (+6 days) weeks of pregnancy (recruitment visit)
  Adiponectine (ug/mL); insulin (ng/mL); C-peptide (ng/mL); leptin (ng/mL); resistin (ng/mL)
Abdominal Fat Thickness | Between 11 (+0 days) and 13 (+6 days) weeks of pregnancy (recruitment visit)
  Ultrasound evaluation, measures expressed in mm. Abdominal Subcutaneous Fat Thickness (ASFT): lower ASFT (thickness of ASFT at the intersection of the horizontal line between the highest points of the iliac crest and the alba line, measuring the thickness of the external face of the rectus abdominis muscle at the skin's surface, with the minimum possible pressure applied on the skin); upper ASFT (subcutaneous adipose thickness at the maximum vertical distance from the skin line to the anterior edge of the linea alba, after a mid-sagittal section of the upper maternal abdomen, with the minimum possible pressure from the probe).
  Visceral Abdominal Fat Thickness (VAT): adipose tissue in the anterior abdomen at the xipho-umbilical line.
Fetal Adipose Tissue Deposits | Between 28 (+0 days) and 40 (+6 days) weeks of pregnancy (third trimester control visit)
  Ultrasound evaluation, measures expressed in mm. Thickness of subcutaneous adipose tissue in the abdomen, thigh, arm.

SECONDARY OUTCOMES:
Gestational diabetes prevalence | Between 14 (+0 days) and 27 (+6 days) weeks of pregnancy (second trimester control visit) and third trimester control visit
  Prevalence of gestational diabetes according to the class of risk (high or low risk)
Obstetric complications and mode of delivery | Recruitment visit; second trimester control visit; third trimester control visit; in the day of the delivery, in average 6 months after recruitment visit (post-partum visit)
  Occurrence of gestational hypertension, pre-eclampsia, intrauterine growth restriction, preterm labour. Mode of delivery (spontaneous, cesarean section, operative).

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Simoncini, MD. PhD., Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No